CLINICAL TRIAL: NCT02031770
Title: Effect of Treatment of Metabolic Acidosis on Vascular Function in Patients With Chronic Kidney Disease: A Pilot Study
Brief Title: Metabolic Acidosis and Vascular Function in Patients With Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Denver Health and Hospital Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13-2017
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Results first posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Metabolic Acidosis; Chronic Kidney Disease
Keywords: vascular endothelial cells
MeSH Terms: conditions — Acidosis; Renal Insufficiency, Chronic | interventions — Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Treatment/Control (Other): Patients will start with sodium bicarbonate treatment then switch to control (no treatment)
  Interventions: Drug: Sodium bicarbonate; Other: Control
- B: Control/Treatment (Other): Patients will start with control (no treatment) then switch to sodium bicarbonate treatment
  Interventions: Drug: Sodium bicarbonate; Other: Control

INTERVENTIONS:
Drug: Sodium bicarbonate — Subjects will be treated with oral sodium bicarbonate two to three times per day for a goal serum bicarbonate (HCO3-) of ≥ 23 meq/L.
Other: Control — subjects will receive no treatment

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death in patients with chronic kidney disease (CKD) and large artery damage is a major factor that contributes to death. Metabolic acidosis is a common complication of CKD resulting from an inability of the diseased kidney to excrete the daily dietary acid load and it is associated with all-cause mortality in patients with CKD. However, the effect of treatment of metabolic acidosis with oral sodium bicarbonate on endothelial dysfunction and arterial stiffness in patients with CKD has not been evaluated. The investigators propose a prospective, randomized, controlled, open-label 14-week crossover pilot study examining the effect of treatment of metabolic acidosis with oral sodium bicarbonate on vascular endothelial function in 20 patients with CKD stage IV with metabolic acidosis.

ELIGIBILITY:
Inclusion Criteria

* Age 40-70 years
* CKD stage IV (eGFR 15-29 ml/min/1.73m2; stable renal function in the past 3 months)
* Serum bicarbonate level of < 20 and ≥ 16 meq/L (at least 2 consecutive weekly measurements)
* Body mass index < 40 kg/m2 (FMD measurements can be inaccurate in severely obese patients)
* Ability to give informed consent
* Stable anti-hypertensive, diabetic and lipid lowering regimen for at least one month prior to randomization

Exclusion Criteria:

* Significant comorbid conditions that lead the investigator to conclude that life expectancy is less than 1 year
* Uncontrolled hypertension
* Expected to undergo living related kidney transplant in next 6 months
* Expected to start dialysis in next 3 months
* Overt congestive heart failure
* Use of sevelamer
* Use of calcium carbonate

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Kendrick, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | A: Treatment/Control | B: Control/Treatment
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Study Participants: Patients will start with sodium bicarbonate treatment then switch to control (no treatment)
  Sodium bicarbonate: Subjects will be treated with oral sodium bicarbonate two to three times per day for a goal serum bicarbonate (HCO3-) of ≥ 23 meq/L.
  Control: subjects will receive no treatment
Arm/Group | Study Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Brachial Artery Flow Mediated Dilation (FMD)
Description: The primary endpoint is change in brachial artery FMD between treatment and control conditions. Each treatment period is 6 weeks in duration with a 2 week washout period in between. Outcome measures will be repeated at the beginning and end of each period.
Time Frame: 6 weeks and 12 weeks
Measure: Mean (Standard Deviation); unit: absolute change in percent FMD
Arm/Group | Treatment | Control
Number analyzed (Participants) | 20 | 20
absolute change in percent FMD | 1.1 (2.6) | -0.7 (1.9)

ADVERSE EVENTS:
Arm/Group | Treatment | Control
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 11/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=20) | Control (N=20)
Nausea (Gastrointestinal disorders) | 7 (7) | 0 (0)
Leg swelling (Cardiac disorders) | 4 (4) | 0 (0) — lower extremity edema

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes